CLINICAL TRIAL: NCT02656589
Title: A Perspective Study of the Predictive Value of microRNA in Patients With HER2 Positive Advanced Stage Breast Cancer Who Were Treated With Herceptin
Brief Title: microRNA of Human Epidermal Growth Factor Receptor 2 （HER2）Positive Patient Treated With Herceptin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other); Huiping Li,M.D., Ph.D.,Peking University Cancer Hospital (Unknown)
Responsible Party: Principal Investigator, Erwei Song, M.D., Ph.D., President of Sun Yat-Sen Memorial Hospital, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SSC201512
Record Dates: First submitted 2016-01-08; First posted 2016-01-15 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; herceptin; microRNA
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Herceptin probable sensitive group: Plasma microRNAs will be collected using microRNA extraction kit according to manufacturer's instructions; and their expression levels are analyzed by quantitative polymerase chain reaction (qPCR).According to microRNAs - herceptin predictive model(reported by our team), the patients will be considered as Herceptin probable sensitive group
  Interventions: Drug: Capecitabine; Drug: Trastuzumab
- Herceptin probable resistant group: Plasma microRNAs will be collected using microRNA extraction kit according to manufacturer's instructions; and their expression levels are analyzed by quantitative polymerase chain reaction (qPCR).According to microRNAs - herceptin predictive model(reported by our team), the patients will be considered as Herceptin probable resistant group
  Interventions: Drug: Capecitabine; Drug: Trastuzumab

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will be administered orally at a dose of 2500mg/m2 daily for 3 months (Day 1 to 14 of a 21-day cycle)
  Other Names: Xeloda
Drug: Trastuzumab — patients will receive herceptin intravenous infusion at a dose of 6mg on day 1 of each cycle
  Other Names: Herceptin

SUMMARY:
This projective observational study is planned to enroll more than 300 advanced breast cancer patients, who were proved as Her-2 positive using fluorescence in situ hybridization (FISH) and / or immunohistochemistry, and 100 healthy donors as control. Before treatment, the plasma microRNA will be collected and detected by microRNA extraction kit and quantitative polymerase chain reaction (qPCR), respectively. After analyzed their microRNA expression by microRNA predictive model, previously reported by our team, all of enrolled patients will be classified as "probable sensitive group" or "probable resistant group". Herceptin combined with other chemotherapy will be the backbone of salvage treatment and used for at least 3 months; the change of local masses and metastasis lesions after treatment will be documented to evaluate the response. Based on these results, investigator aim to construct a mathematical predictive model by analyzing the correlation of baseline microRNA expression level and the prognosis of patients. And a diagnosis microRNA kit will be planned and manufactured

ELIGIBILITY:
Inclusion Criteria:

1. The patients signed the written informed consent
2. female patient who is ≥ 18yrs,
3. HER2 positive: immunohistochemistry (+++) or FISH (+)
4. stage IV
5. the patients have no history of chemotherapy ,hormone therapy,radiotherapy or surgery after diagnosis of breast cancer
6. the result of patients' blood tests are as follow: WBC≥3.0×109/L; Plt≥100×109/L;AST/SGOT or ALT/AGPT≤tripple of normal upper limit; Creatinine<double of the normal upper limit
7. ECOG scores are 0 or 1 .
8. The patient is able to take oral pills

Exclusion Criteria:

1. The patient was never exposed to herceptin.
2. The patient suffered from other non-breast malignancy in the last 5 years, except for cervical carcinoma in situ, radical basal cell carcinoma or squamous cell carcinoma.
3. The life expectancy is less than 3 months.
4. Severe hepatic function disorder, Child Pugh grade C.
5. Severe cardiac function disorder, cardiac function is more than grade III;
6. Prolonged QT interval;
7. Arrhythmia or taking anti-arrhythmia drugs;
8. Pregnant or breast feeding female.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced breast cancer patients first diagnosis in Sun Yat-sen Memorial Hospital, Sun Yat-sen University. Informed consent must be obtained for all of the included patients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival of patients | progression free survival (PFS) was defined as the interval from the diagnosis of advanced breast cancer with HER2 positive to disease progression, relapse, death due to any causes or last follow-up.The follow-up interval is 2 years.
overall survival of patients | Overall survival was defined as the interval from the diagnosis of advanced breast cancer with HER2 positive to death due to any causes or last follow-up,The follow-up interval is 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, Ph.D, Study Chair — Sun Yat-Sen Memerial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Hur K, Toiyama Y, Schetter AJ, Okugawa Y, Harris CC, Boland CR, Goel A. Identification of a metastasis-specific MicroRNA signature in human colorectal cancer. J Natl Cancer Inst. 2015 Feb 6;107(3):dju492. doi: 10.1093/jnci/dju492. Print 2015 Mar. PMID 25663689
- [Result] Jiang L, Cheng Q, Zhang BH, Zhang MZ. Circulating microRNAs as biomarkers in hepatocellular carcinoma screening: a validation set from China. Medicine (Baltimore). 2015 Mar;94(10):e603. doi: 10.1097/MD.0000000000000603. PMID 25761179
- [Result] Kleivi Sahlberg K, Bottai G, Naume B, Burwinkel B, Calin GA, Borresen-Dale AL, Santarpia L. A serum microRNA signature predicts tumor relapse and survival in triple-negative breast cancer patients. Clin Cancer Res. 2015 Mar 1;21(5):1207-14. doi: 10.1158/1078-0432.CCR-14-2011. Epub 2014 Dec 29. PMID 25547678
- [Result] Xiang M, Zeng Y, Yang R, Xu H, Chen Z, Zhong J, Xie H, Xu Y, Zeng X. U6 is not a suitable endogenous control for the quantification of circulating microRNAs. Biochem Biophys Res Commun. 2014 Nov 7;454(1):210-4. doi: 10.1016/j.bbrc.2014.10.064. Epub 2014 Oct 18. PMID 25450382
- [Result] Zhai R, Wei Y, Su L, Liu G, Kulke MH, Wain JC, Christiani DC. Whole-miRNome profiling identifies prognostic serum miRNAs in esophageal adenocarcinoma: the influence of Helicobacter pylori infection status. Carcinogenesis. 2015 Jan;36(1):87-93. doi: 10.1093/carcin/bgu228. Epub 2014 Nov 8. PMID 25381453
- [Result] Gururajan M, Josson S, Chu GC, Lu CL, Lu YT, Haga CL, Zhau HE, Liu C, Lichterman J, Duan P, Posadas EM, Chung LW. miR-154* and miR-379 in the DLK1-DIO3 microRNA mega-cluster regulate epithelial to mesenchymal transition and bone metastasis of prostate cancer. Clin Cancer Res. 2014 Dec 15;20(24):6559-69. doi: 10.1158/1078-0432.CCR-14-1784. Epub 2014 Oct 16. PMID 25324143
- [Result] Parpart S, Roessler S, Dong F, Rao V, Takai A, Ji J, Qin LX, Ye QH, Jia HL, Tang ZY, Wang XW. Modulation of miR-29 expression by alpha-fetoprotein is linked to the hepatocellular carcinoma epigenome. Hepatology. 2014 Sep;60(3):872-83. doi: 10.1002/hep.27200. Epub 2014 Jul 25. PMID 24798303
- [Result] Masuda S, Izpisua Belmonte JC. Re: Serum miR-21 as a diagnostic and prognostic biomarker in colorectal cancer. J Natl Cancer Inst. 2014 Mar;106(3):djt457. doi: 10.1093/jnci/djt457. Epub 2014 Mar 1. No abstract available. PMID 24586105
- [Result] Schwarzenbach H, Nishida N, Calin GA, Pantel K. Clinical relevance of circulating cell-free microRNAs in cancer. Nat Rev Clin Oncol. 2014 Mar;11(3):145-56. doi: 10.1038/nrclinonc.2014.5. Epub 2014 Feb 4. PMID 24492836
- [Result] Chan M, Liaw CS, Ji SM, Tan HH, Wong CY, Thike AA, Tan PH, Ho GH, Lee AS. Identification of circulating microRNA signatures for breast cancer detection. Clin Cancer Res. 2013 Aug 15;19(16):4477-87. doi: 10.1158/1078-0432.CCR-12-3401. Epub 2013 Jun 24. PMID 23797906
- [Result] Wang Y, Gu J, Roth JA, Hildebrandt MA, Lippman SM, Ye Y, Minna JD, Wu X. Pathway-based serum microRNA profiling and survival in patients with advanced stage non-small cell lung cancer. Cancer Res. 2013 Aug 1;73(15):4801-9. doi: 10.1158/0008-5472.CAN-12-3273. Epub 2013 Jun 17. PMID 23774211
- [Result] Li A, Yu J, Kim H, Wolfgang CL, Canto MI, Hruban RH, Goggins M. Serum miR-1290 as a marker of pancreatic cancer--response. Clin Cancer Res. 2013 Sep 15;19(18):5252-3. doi: 10.1158/1078-0432.CCR-13-1899. Epub 2013 Jul 23. No abstract available. PMID 23881921
- [Result] van Schooneveld E, Wouters MC, Van der Auwera I, Peeters DJ, Wildiers H, Van Dam PA, Vergote I, Vermeulen PB, Dirix LY, Van Laere SJ. Expression profiling of cancerous and normal breast tissues identifies microRNAs that are differentially expressed in serum from patients with (metastatic) breast cancer and healthy volunteers. Breast Cancer Res. 2012 Feb 21;14(1):R34. doi: 10.1186/bcr3127. PMID 22353773
- [Result] Jackson DB. Serum-based microRNAs: are we blinded by potential? Proc Natl Acad Sci U S A. 2009 Jan 6;106(1):E5. doi: 10.1073/pnas.0809999106. Epub 2008 Dec 23. No abstract available. PMID 19106287
- [Result] Roth C, Rack B, Muller V, Janni W, Pantel K, Schwarzenbach H. Circulating microRNAs as blood-based markers for patients with primary and metastatic breast cancer. Breast Cancer Res. 2010;12(6):R90. doi: 10.1186/bcr2766. Epub 2010 Nov 3. PMID 21047409
- [Result] Li LM, Hu ZB, Zhou ZX, Chen X, Liu FY, Zhang JF, Shen HB, Zhang CY, Zen K. Serum microRNA profiles serve as novel biomarkers for HBV infection and diagnosis of HBV-positive hepatocarcinoma. Cancer Res. 2010 Dec 1;70(23):9798-807. doi: 10.1158/0008-5472.CAN-10-1001. Epub 2010 Nov 23. PMID 21098710
- [Result] Li J, Wang Y, Yu W, Chen J, Luo J. Expression of serum miR-221 in human hepatocellular carcinoma and its prognostic significance. Biochem Biophys Res Commun. 2011 Mar 4;406(1):70-3. doi: 10.1016/j.bbrc.2011.01.111. Epub 2011 Feb 3. PMID 21295551